CLINICAL TRIAL: NCT04195048
Title: Mechanism and Outcome of Acute Ischemic Stroke in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 9
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke; Cancer
Keywords: Ischemic Stroke, Cancer
MeSH Terms: conditions — Ischemic Stroke; Neoplasms | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients with acute ischemic stroke: Eighty patients previously or currently suffering from manifest cancer on or not on cancer treatment who developed stroke
  Interventions: Other: Risk factors
- Control patients with acute ischemic stroke without cancer: Eighty patients with acute ischemic stroke without cancer
  Interventions: Other: Risk factors

INTERVENTIONS:
Other: Risk factors — Risk factors: modifiable and unmodifiable risk factors

SUMMARY:
Stroke is a part of circulatory diseases which are the primary cause of death in Egypt. It accounts 14% of all deaths thus ranks the 2nd after ischemic heart disease. Cancer accounts 9% of population mortality in Egypt. Nearly 108,600 Egyptians newly diagnosed with cancer each year. The interrelationship between stroke and cancer is complex. Cancer may directly or indirectly lead to stroke via: hypercoagulability, nonbacterial thrombotic endocarditis (NBTE), direct tumor compression of blood vessels or treatment-related effects which potentiate stroke.

The risk of ischemic stroke after chemotherapy is largely increased by the use of certain types of chemotherapy not only by cancer histologic type. Brain infarction usually a subsequent complication appears sometimes shortly after chemotherapy. Chronic radiation vasculopathy that affects medium and large intra- and extra-cranial arteries is characterized by increasing rates of hemodynamic significant stenosis with time after radiotherapy.

The study aims to clarify the relation between cancer and its treatment with ischemic stroke by discussing the different mechanisms by which a vascular insult happen causing neurological deficit. The study provides more information about cancer patients with higher risk to develop ischemic stroke more than other patients by identifying co morbidities and dosage of cancer treatment that causes cerebrovascular insults.

DETAILED DESCRIPTION:
* Retrospective study was conducted on patients diagnosed with cancer receiving chemotherapy or radiotherapy to evaluate the relation between cancer or cancer therapies and ischemic stroke development.
* Patients had been recruited from the oncology center, nuclear medicine department and neurology department in Mansoura University and private centers.

After obtaining informed consent, patients are subjected to the following:

1. Detailed History taking of previous cerebrovascular insults and cancer diagnosis onset and therapies.
2. Determination of major cerebrovascular risk factors as :

   * Hypertension: which is diagnosed when a patient had received antihypertensive treatment or when hypertension is diagnosed during the hospital stay by repeated detection of blood pressure of 140/90 mm Hg .
   * Diabetes mellitus (DM): diagnosis based on history of DM with or without current treatment or random blood glucose is 200mg/dl or higher.
   * Hypercholesterolemia: diagnosis based on history of hypercholesterolemia with current treatment or serum cholesterol level >220mg/dl.
   * Smoking: is coded when the patient is a current smoker or an ex-smoker within 5 years.
   * Cardiac abnormality
3. Physical and neurological examination.
4. Investigations:

   * Laboratory investigations as complete blood count, lipid profile, coagulation profile, CRP , D dimer .
   * Radiological investigations: MRI brain to detect vascular abnormalities that may be associated with cancer such as: lacunar infarction , white matter changes and microbleeds.
5. For all patients in the prospective group the duration and type of chemotherapy, dose of radiotherapy was recorded.

ELIGIBILITY:
Inclusion Criteria:

* 80 patients previously or currently suffering from manifest cancer on or not on cancer treatment who developed stroke
* 80 control patient with ischemic storke without cancer

Exclusion Criteria:

* Patients developed cerebrovascular insults prior to the onset of cancer
* Cancer patients with symptoms mimic stroke.
* Cancer patients with focal neurological deficit due to direct effect of malignant tumor.
* Patients missed their follow up.
* Patients with traditional cerebrovascular risk factors such as (hypertension, hyperlipidemia, diabetes and atrial fibrillation) prior to cancer diagnosis.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Retrospective study was conducted on patients diagnosed with cancer receiving chemotherapy or radiotherapy to evaluate the relation between cancer or cancer therapies and ischemic stroke development.
  * Patients had been recruited from the oncology center, nuclear medicine department and neurology department in Mansoura University and private centers.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 6 months
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No